CLINICAL TRIAL: NCT01345071
Title: PreConceptional Counselling in Active Rheumatoid Arthritis
Acronym: PreCARA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: J.M.W. Hazes (Other)
Collaborators: Erasmus Medical Center (Other); Dutch Arthritis Association (Industry)
Responsible Party: Sponsor-Investigator, J.M.W. Hazes, Head of the Department, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: ErasmusMC-MEC-2011-032
Record Dates: First submitted 2011-04-13; First posted 2011-04-29 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis; Pregnancy
Keywords: Rheumatoid Arthritis; Pregnancy; Anti-TNF; Preconceptional counselling; Disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood of mother before, during and after pregnancy; cordblood of newborn; blood of newborn if anti-TNF in cord blood was above reference level.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients: RA patients with active disease or current use of anti-TNF. Treatment is according to treat to target principles.

SUMMARY:
The first objective of the study is to evaluate a treat to target treatment strategy in women with moderate to high disease activity of RA and a pregnancy wish, from pre-pregnancy. The treatment strategy is based on deliberate treatment decisions to lower disease activity, including the continuation or start of biological treatment (in particular anti-Tumor Necrosis Factor [anti-TNF]), based on a standard care protocol in the Erasmus MC. The second objective is to evaluate the safety of the use of anti-TNF during pregnancy among women with a rheumatic disease that require the use of anti-TNF before or during pregnancy.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is an auto-inflammatory disease that particularly involves chronic inflammation of the joints.The disease is in essence a systemically active one that can affect almost any organ. Pregnancy can spontaneously reduce the activity of RA. This phenomenon has been investigated in the PARA-study (Pregnancy-induced Amelioration of Rheumatoid Arthritis study), a nationwide prospective cohort study initiated and coordinated by the department of Rheumatology, Erasmus University Medical Center, Rotterdam the Netherlands.

The PARA-study reconfirmed previous data that RA improved during pregnancy. However, it also showed that this improvement was less pronounced than previously thought since > 50% of RA-patients still had active disease during third trimester of pregnancy. It also demonstrated that active RA was associated with lower birth weight and that children of mothers with active RA demonstrated rapid catch up growth in weight. Lower birth weight as well as rapid catch up growth in weight have been shown to be associated with a less favorable cardiovascular profile in early adulthood. Finally, it showed that time to pregnancy is prolonged in RA-patients with active disease. Also the use of prednisone > 7,5 mg daily or the use of NSAIDs (Non-Steroidal Anti-Inflammatory Drugs) were associated with a prolonged time to pregnancy. These latter associations were independent of disease activity.

The findings of the PARA-study implicate that one should strive for low disease activity in women with RA and a pregnancy wish, but that in the meantime NSAIDs and doses of prednisone exceeding 7.5 mg daily should be avoided. Since common drugs to treat RA, like methotrexate, are incompatible with pregnancy, lowering disease activity in pregnant RA-patients or with a pregnancy wish becomes a real challenge for the patient and the treating physician. This all underscores the importance of new treatment modalities for RA-patients with a pregnancy wish.

In the last decade new treatment options for RA, the so-called biologicals, became available. During pregnancy the most experience has been gained with biologicals belonging to the class of anti-TNF therapy. In the USA, anti-TNF has been approved for use during pregnancy as a FDA (Food and Drug Administration) class B (i.e. Animal reproduction studies fail to demonstrate a risk to the fetus, and adequate, but well-controlled, studies of pregnant women have not been conducted). Registry studies show that anti-TNF use seems to be safe during pregnancy in humans also. Furthermore, anti-TNF therapy has been used intentionally preconceptionally to improve the chance of pregnancies in women with recurrent spontaneous abortions. Since no randomized controlled trials can be done during pregnancy, circumstantial evidence has led to decision making in daily practice. In case of high disease activity use of anti-TNF to control disease activity outweighs the risk of potential harm to the foetus.

Most anti-TNF medications are monoclonal antibodies of the IgG class. For that reason these antibodies are, from around week 14 of gestation, actively transported across the placenta. When used into third trimester of pregnancy, higher levels of these TNF-alpha antibodies are reached in the fetal circulation compared to the maternal circulation, making the newborn more prone for infections. Vaccination of newborns with live inactivated vaccines are therefore contraindicated till anti-TNF alpha antibody levels are not detectable anymore. It is often advised to stop anti-TNF in the first trimester of pregnancy. The rationale behind this approach is that RA improves during pregnancy anyway and that it is safe to taper off medication. In addition it is thought that with discontinuation of anti-TNFearly during pregnancy no placental transfer of anti-TNF antibodies will take place. However, currently no scientific evidence is available to support both assumptions.

An alternative approach is to prescribe Certolizumab during pregnancy or in women with a pregnancy wish. Certolizumab is a pegylated antibody against TNF-alpha. Since it lacks an Fc-tail it is not transported across the placenta and only trace amounts can be detected in the newborn. In the Erasmus MC a protocol was recently developed to standardize care for patients (already pregnant or with a pregnancy wish) that in theory might benefit from treatment with anti-TNF therapy. This protocol is being evaluated in the Pre-CARA study.

The Pre-CARA study is a continuation of the previous PARA study, but focuses on RA patients with high disease activity and a pregnancy wish. The first objective is to evaluate a treat to target treatment strategy in women with moderate to high disease activity of RA and a pregnancy wish, from pre-pregnancy till six months after delivery. The treatment strategy is based on deliberate treatment decisions to lower disease activity, including the continuation or start of biological treatment (anti-TNF), based on a standard care protocol in the Erasmus MC. The second objective is to evaluate the safety of the use of anti-TNF during in women with any chronic arthritide who require the use of this medication preconceptionally and/or during pregnancy.

ELIGIBILITY:
Inclusion criteria for first objective (150 subjects)

* Rheumatoid Arthritis according to 2010 ACR/EULAR criteria
* active pregnancy wish
* either DAS28(3)CRP > 3.2 or the current use of anti-TNF

Inclusion criteria for second objective (no limit on number of subjects needed, recruitment will end when 150 RA patients have been included)

* rheumatic disease that requires the use of anti-TNF before or during pregnancy
* active pregnancy wish

Exclusion criteria:

- none

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: For first objective: Women with high disease activity of RA and a pregnancy wish.
  For second objective: Women with a rheumatic disease that requires the use of anti-TNF before or during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2021-06 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
DAS28(3)CRP at all study points | Every 3 months from baseline till 6 months after delivery

SECONDARY OUTCOMES:
Time to pregnancy | At baseline and every 3 months till pregnant
  Patient is asked whether is she is pregnant. Pregnancy is defined as positive pregnancy test or ultrasound.
Number of miscarriages | After conception, every 3 months
  Patients normally report miscarriages spontaneously at the next visit after miscarriage or contact the research nurse themselves to report this. If not, and patient is not pregnant anymore, reason for ending of pregnancy will be asked.
Complications during pregnancy | Every 3 months during pregnancy and first visit after delivery
  Complications are: hypertensive disorders, pre-eclampsia, diabetes, mode of delivery, hospitalization
Gestational age of child | First visit after delivery
Birth weight of child | First visit after delivery
Congenital malformations | First visit after delivery
Growth of child and tempo of growth during first year | One year after birth
Maternal serum levels of anti-TNF | Every three months during pregnancy
Levels of anti-TNF in cord blood | Collected at birth
Levels of anti-TNF in child | Every six weeks after birth
  Only if anti-TNF in cord blood was above reference value, blood will be drawn from the newborn every six weeks, till anti-TNF-levels are below reference value

CONTACTS AND LOCATIONS:
Overall Officials: Radboud Dolhain, PhD MD, Principal Investigator — Staff Rheumatologist
Locations (1):
- ErasmusMC, University Medical Center Rotterdam, dept. of Rheumatology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
This will be discussed in the research group

REFERENCES:
- [Background] de Man YA, Dolhain RJ, Hazes JM. Disease activity or remission of rheumatoid arthritis before, during and following pregnancy. Curr Opin Rheumatol. 2014 May;26(3):329-33. doi: 10.1097/BOR.0000000000000045. PMID 24614279
- [Background] de Man YA, Dolhain RJ, van de Geijn FE, Willemsen SP, Hazes JM. Disease activity of rheumatoid arthritis during pregnancy: results from a nationwide prospective study. Arthritis Rheum. 2008 Sep 15;59(9):1241-8. doi: 10.1002/art.24003. PMID 18759316
- [Background] de Man YA, Hazes JM, van der Heide H, Willemsen SP, de Groot CJ, Steegers EA, Dolhain RJ. Association of higher rheumatoid arthritis disease activity during pregnancy with lower birth weight: results of a national prospective study. Arthritis Rheum. 2009 Nov;60(11):3196-206. doi: 10.1002/art.24914. PMID 19877045
- [Derived] Quaak CH, Kluivers ACM, Baart SJ, Smeele HTW, Neuman RI, Saleh L, Visser W, Danser AHJ, Dolhain RJEM. Tumor Necrosis Factor Inhibitor Use Increases Birthweight in Pregnant Women With Rheumatoid Arthritis Independently of the Soluble Fms-Like Tyrosine Kinase-1/Placental Growth Factor Ratio. J Am Heart Assoc. 2024 Apr 2;13(7):e032655. doi: 10.1161/JAHA.123.032655. Epub 2024 Mar 27. PMID 38533985